CLINICAL TRIAL: NCT02312856
Title: Adjunctive Neurovascular Support for Wide-neck Aneurysm Embolization and
Brief Title: Adjunctive Neurovascular Support for Wide-neck Aneurysm Embolization and Reconstruction
Acronym: ANSWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulsar Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0014
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PulseRider aneurysm (Experimental): Endovascular treatment of intracranial aneurysms
  Interventions: Device: PulseRider

INTERVENTIONS:
Device: PulseRider — Adjunctive device for endovascular embolization of intracranial aneurysms

SUMMARY:
This study is designed to evaluate the safety of the PulseRider in patients undergoing treatment for bifurcation basilar or carotid terminus aneurysms.

DETAILED DESCRIPTION:
Primary Endpoints:

* Safety: Death or stroke in downstream territory to 180-days post-procedure
* Technical Success: Device placement success and ability to retain coils at the time of the index procedure
* Rate of aneurysm occlusion at Day zero (0) and 180 days

Additional Evaluations to 180-days and at 365-day follow up:

* Rate of aneurysm occlusion at 365 days
* Device movement or migration
* Stenosis
* Rate of incidence of new neurological deficits
* Complication rate (neurological and non-neurological)

ELIGIBILITY:
Inclusion Criteria:

* Patient who presents with an angiographically confirmed, wide neck intracranial aneurysms located at a bifurcation of the basilar artery or carotid terminus artery
* The target aneurysm is in a vessel with a diameter of 2.7 mm to 4.5 mm.
* The patient is 18 years or older at the time of consent
* The patient has signed the IRB/EC approved informed consent form
* In the opinion of the physician, placement of the PulseRider is technically feasible and clinically indicated
* Subject has mental capacity and is willing and able to comply with protocol requirements and follow-up

Exclusion Criteria:

* Unstable neurological deficit (condition worsening within the last 90 days)
* Subarachnoid Hemorrhage (SAH) within the last 60 days
* Irreversible bleeding disorder
* mRS score ≥3
* Patient has another aneurysm which, in the Investigator's opinion, will require treatment within the follow up period (365 days)
* Platelet count < 100 x 103 cells/mm3
* Inability to tolerate, adverse reaction or contraindication to taking aspirin or clopidogrel
* A history of contrast allergy that cannot be medically controlled
* Known allergy to nickel
* Relative contraindication to angiography (e.g., serum creatinine > 2.5 mg/dL)
* Woman with child-bearing potential who cannot provide a negative pregnancy test
* Evidence of active infection
* Other conditions of the heart, blood, brain or intracranial vessels that carry a high risk of neurologic events
* Evidence of disease or condition expected to compromise survival or ability to complete follow-up assessments during the 365-day follow-up period
* Extracranial stenosis greater than 50% in the parent artery requiring access to the lesion
* Intracranial stenosis greater than 50% in the treated vessel
* Extreme vessel tortuosity that prohibits appropriate control of the micro-guide wire and/or the PulseRider delivery wire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2015-10-13 (Actual); Study Completion 2016-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Spiotta, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PulseRider: Subjects 1 year Follow Up
Period: Overall Study
Arm/Group | PulseRider
Started (10/22/2014) | 34
Completed (11/07/2015) | 30
Not Completed | 4
Not completed — Death | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Male and female subjects, ≥18 years of age with a wide neck (≥ 4 mm or dome to neck ratio < 2) basilar or carotid terminus aneurysm located at a bifurcation. Subjects with acutely ruptured aneurysms were excluded from the study. The aneurysm parent vessel measurements were required to be between 2.7 mm and 4.5 mm to be suitable for the procedure.
Groups:
- PulseRider: Total Participants
Arm/Group | PulseRider
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: year]
  Age | 60.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Raymond Score I/II or Experienced Neurological Death
Description: Raymond Scale- an angiographic classification scheme for grading the occlusion of endovascularly treated intracranial aneurysms. Achieving a Raymond Score I/II.
  class I: complete obliteration class II: residual neck class III: residual aneurysm class IIIa: contrast opacification within the coil interstices of a residual aneurysm class IIIb: contrast opacification outside the coil interstices, along the residual aneurysm wall. Raymond I is typically associated with better outcomes. The primary outcome of the study looked at safety (death or stroke) and Rate of Aneurysm occlusion (assess by Raymond Roy scores) the two are different. The RR Score is an assessment of occlusion and not used to assess death.
Time Frame: 180 days post procedure
Population: One enrolled participant had MRA performed instead of an angiogram and is excluded from Raymond Score analysis.
Measure: Number; unit: Participants
Groups:
- Safety: Number of affected participants
Arm/Group | Safety
Number analyzed (Participants) | 34
Participants
  # participants experienced Neurological Death | 0
  # participants who scored Raymond Score I/II: number analyzed (Participants) | 33
  # participants who scored Raymond Score I/II | 29

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from enrollment of the first subject through 1 year for all subjects.
Description: All AEs and SAEs were included in the reports to FDA throughout the study.
Groups:
- Number: Number of Participants between the procedure and 365 days
Arm/Group | Number
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 12/34
Other Adverse Events (participants affected / at risk) | 27/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Number (N=34)
Death (Cardiac disorders) | 1 (1)
Stroke (Cardiac disorders) | 5 (5)
Cauda Equina Syndrome (Nervous system disorders) | 1 (1)
Coil perforation of aneurysm (Surgical and medical procedures) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Possible seizure (Nervous system disorders) | 1 (1)
Leg Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Right or left side weakness
Femoral Occlusion (Vascular disorders) | 1 (1)
Hypotension (Blood and lymphatic system disorders) | 1 (1) — Hypotension
OTHER ADVERSE EVENTS (reported when occurring in more than 2.9% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Number (N=34)
Headache (Vascular disorders) | 10 (10)
Depression (Psychiatric disorders) | 2 (2)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (General disorders) | 4 (4)
Constipation (General disorders) | 2 (2)
Ecchymosis (General disorders) | 2 (2)
Hematoma (General disorders) | 2 (2)
Dizziness (General disorders) | 1 (1)
Respiratory problems (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Nose Bleed (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days